CLINICAL TRIAL: NCT07279987
Title: Comparison of Combined Rotational Atherectomy With Intravascular Lithotripsy Versus Super-High Pressure Balloon Angioplasty for Heavily Calcified Coronary Lesions (CRUSH-CALC Study)
Brief Title: Comparison of RA-IVL and RA-SHP in Calcified Coronary Lesions
Acronym: CRUSH-CALC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lin Zhao (Other)
Collaborators: China-Japan Friendship Hospital (Other); Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Lin Zhao, Cheif of Cardiovascular department, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-ke-874
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Vascular Calcification
Keywords: Coronary Artery Disease; Percutaneous Coronary Intervention; Vascular calcification; Rotational atherectomy; Intravascular lithotripsy; Super high-pressure balloon; Major adverse cardiovascular events; Plaque modification
MeSH Terms: conditions — Vascular Calcification; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotational Atherectomy + Super High-Pressure Balloon (Experimental): Patients with severely calcified coronary lesions undergo rotational atherectomy followed by super high-pressure balloon angioplasty (SHPB) for calcium modification, then drug-eluting stent implantation with intravascular imaging guidance
  Interventions: Device: Super High-Pressure Non-Compliant Balloon
- Rotational Atherectomy + Intravascular Lithotripsy (Active Comparator): Patients with severely calcified coronary lesions undergo rotational atherectomy followed by intravascular lithotripsy (IVL) for calcium modification, then drug-eluting stent implantation with intravascular imaging guidance
  Interventions: Device: Intravascular Lithotripsy System

INTERVENTIONS:
Device: Super High-Pressure Non-Compliant Balloon — The super high-pressure balloon is a non-compliant balloon catheter capable of withstanding inflation pressures up to 35-40 atmospheres. The balloon is sized 1:1 to the reference vessel diameter and positioned across the calcified lesion. Inflation follows a stepwise pressure escalation protocol: 12 atm → 20 atm → 25 atm → 30 atm → 35 atm, with each pressure level maintained for 10-20 seconds. The high-pressure inflation creates controlled fractures in calcified plaque to facilitate subsequent stent deployment and expansion. The device is specifically designed for modification of severely calcified coronary lesions.
  Other Names: SHPB; Ultra-High Pressure Balloon; Non-Compliant Balloon (rated to 35-40 atm); OPN NC Balloon
  Arms: Rotational Atherectomy + Super High-Pressure Balloon
Device: Intravascular Lithotripsy System — The intravascular lithotripsy (IVL) system is a balloon-based catheter device that delivers sonic pressure waves to fracture calcium in coronary arteries. The IVL balloon is sized 1:1 to the reference vessel diameter and positioned across the calcified lesion. Once inflated to 4 atm, the system delivers up to 80 pulses of localized pulsatile mechanical energy (50 Hz) to create circumferential and longitudinal calcium fractures in both superficial and deep calcium layers. Each treatment cycle consists of 10 pulses over 10 seconds. The device is specifically designed to modify severe coronary calcification to facilitate stent delivery and expansion.
  Other Names: IVL; Coronary Intravascular Lithotripsy; Sonic Pressure Wave Lithotripsy; Shockwave Coronary IVL System
  Arms: Rotational Atherectomy + Intravascular Lithotripsy

SUMMARY:
Study Design Prospective, multicenter, single-blind, randomized controlled trial

Hypothesis In patients with severely calcified coronary lesions undergoing rotational atherectomy (Rota), post-rotational lesion optimization using intravascular lithotripsy (IVL) is non-inferior to super high-pressure balloon (SHPB) in terms of final minimal lumen diameter (MLD), with potential differences in acute lumen gain, stent expansion, and periprocedural complications.

Inclusion Criteria

* Age ≥ 18 years
* De novo coronary lesions with severe calcification confirmed by angiography (moderate-to-severe calcification) and IVUS (calcification grade ≥2 by Mintz classification, or IVUS cannot pass)
* Target vessel reference diameter 2.5-4.0 mm
* Lesion length ≤ 30 mm suitable for rotational atherectomy
* Clinical evidence of ischemia (stable or unstable angina, or functional ischemia testing)
* Planned rotational atherectomy with residual calcification grade ≥2 post-Rota (burr ≤1.5 mm), or inadequate expansion with 2.5 mm non-compliant balloon at nominal pressure
* Written informed consent provided

Exclusion Criteria

* Acute myocardial infarction within 7 days
* Presence of thrombus, chronic total occlusion (CTO), or in-stent restenosis in target vessel
* Lesion located in coronary artery bypass graft
* Severe heart failure (LVEF < 30%)
* Previous stenting or rotational atherectomy in same target vessel
* Known contrast allergy, active bleeding, severe comorbidity with life expectancy < 12 months
* Pregnancy or lactation
* Participation in other interventional clinical trials

Randomization

After initial rotational atherectomy (burr ≤1.5 mm), eligible patients meeting imaging-defined "need for further lesion optimization" criteria will be randomized 1:1 to:

Rota + IVL group: Intravascular lithotripsy using pulsed ultrasonic energy (up to 80 pulses, 8 cycles) followed by stent implantation Rota + SHPB group: Super high-pressure balloon (≥30 atm) expansion followed by stent implantation Stratification by: Study center, Reference vessel diameter (2.5-3.0 mm vs. >3.0-4.0 mm)

Primary Endpoint Post-procedural minimal lumen diameter (MLD) measured by OCT/IVUS immediately after stent implantation and post-dilation Secondary Endpoints Procedural efficacy: Acute lumen gain, final stent expansion rate, minimal stent area, stent apposition Procedural safety: Periprocedural complications including coronary perforation, dissection, no-reflow/slow flow, acute stent thrombosis Clinical outcomes: MACE (composite of cardiac death, myocardial infarction, target vessel revascularization) at 30 days, 6 months, and 12 months Other outcomes: Major bleeding (BARC ≥2), acute kidney injury (KDIGO criteria), procedure duration, contrast volume, radiation exposure Sample Size Total: 162 patients (81 per group)

In-hospital monitoring until discharge Clinical follow-up at 30 days, 6 months, and 12 months Imaging follow-up (OCT/IVUS) selectively at designated centers as per protocol or clinical indication

Study Centers

Three tertiary hospitals with extensive experience in complex coronary interventions and calcified lesion management:

* Beijing Chaoyang Hospital, Capital Medical University (coordinating center)
* China-Japan Friendship Hospital
* Xinhua Hospital, Shanghai Jiao Tong University School of Medicine

Study Duration January 2026 to December 2028 (3 years)

DETAILED DESCRIPTION:
Severely calcified coronary lesions reduce vessel compliance, limit balloon expansion, and impair optimal stent deployment, leading to higher procedural risk. Rotational atherectomy (Rota) can modify superficial calcium but may be insufficient for deep or circumferential calcium. Intravascular lithotripsy (IVL) and super high-pressure balloon angioplasty (SHPB) are both used for additional calcium modification, but direct comparative evidence in the "post-Rota lesion optimization" setting is limited.

This multicenter, prospective, randomized, single-blind trial compares Rota + IVL versus Rota + SHPB for imaging-defined lesion optimization and periprocedural safety in severely calcified de novo coronary lesions, with clinical follow-up through 12 months.

Study design and sites

* Design: Prospective, multicenter, randomized controlled, single-blind trial; 1:1 allocation.
* Sites: Beijing Chaoyang Hospital, Capital Medical University (coordinating center); China-Japan Friendship Hospital; Xinhua Hospital, Shanghai Jiao Tong University School of Medicine.
* Study period: January 2026 to December 2028.
* Sample size: 162 participants (81 per group).
* Blinding: Operators are not blinded. Imaging analysts and/or (if applicable) endpoint adjudicators are blinded to treatment allocation.

Core workflow (screening to final imaging)

1. Screening and baseline assessment

   * Collect clinical data, angiography, and planned OCT/IVUS when applicable.
   * Peri-procedural medications are administered per guideline-based and institutional practice and documented (antiplatelet therapy, intraprocedural anticoagulation, etc.).
2. Initial rotational atherectomy (all participants)

   * Rota is performed using a standardized approach across sites.
   * Maximum burr size: ≤1.5 mm.
   * Key procedural parameters are recorded (burr size, rotational speed, runs, and any complications and treatments).
3. Post-Rota "randomization trigger" assessment

   * OCT/IVUS and/or a protocol-defined balloon test is used to determine whether additional lesion optimization is needed (e.g., residual calcific constraint/inadequate compliance).
   * Eligible participants meeting trigger criteria are randomized 1:1 to IVL or SHPB.
   * Stratification factors: study site; reference vessel diameter (2.5-3.0 mm vs >3.0-4.0 mm).
4. Randomized lesion optimization and stent implantation Rota + IVL arm

   * An appropriately sized IVL balloon is advanced across the lesion.
   * Lithotripsy is delivered per protocol limits (up to 80 pulses/8 cycles).
   * Repeat treatment and/or balloon resizing under imaging guidance is allowed and fully documented.

   Rota + SHPB arm
   * SHPB dilation is performed to modify the lesion.
   * Target pressure: ≥30 atm (pressure escalation steps, inflation duration, and maximum pressure per protocol; all parameters documented).
   * Repeat inflations and/or balloon exchange are allowed and documented. After randomized optimization, stent implantation and post-dilation are performed under imaging guidance. Devices and parameters are recorded (stent and post-dilation balloon sizes, pressures, number of inflations).
5. Immediate post-procedure imaging assessment (endpoint measurements)

   * OCT/IVUS is performed after stent implantation and final post-dilation.
   * Imaging pullbacks must cover the lesion and proximal/distal reference segments and meet minimum quality criteria.
   * Quantitative analysis follows prespecified definitions (e.g., post-procedural MLD, minimal stent area, stent expansion and apposition metrics).
   * Calcium morphology (arc, length, thickness, distribution) is captured for exploratory correlation and subgroup analyses.

Safety monitoring and quality control

* Periprocedural complications (e.g., perforation, dissection, slow-/no-reflow, acute stent thrombosis) are captured, graded, and reported using prespecified definitions and timelines.
* Data are collected using standardized CRFs and a multicenter database for data capture, follow-up tracking, and quality assurance.
* Monitoring focuses on: eligibility, randomization trigger criteria, key imaging timepoints, major safety events, and follow-up completeness.

Follow-up

* In-hospital monitoring until discharge.
* Clinical follow-up at 30 days, 6 months, and 12 months (clinic visit and/or telephone).
* Collection of clinical events, bleeding and renal outcomes, and resource utilization metrics (procedure time, contrast volume, radiation exposure).
* Imaging follow-up (if specified in the protocol or clinically indicated) may be performed selectively at designated centers.

Statistical considerations (overview)

* A noninferiority framework is used to compare the primary imaging outcome between groups.
* Primary analysis population: intention-to-treat (ITT), with supportive per-protocol (PP) analysis.
* Stratification factors are incorporated in the analysis model. Missing imaging data are handled using prespecified methods with sensitivity analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, able to understand the study purpose and voluntarily sign written informed consent
* Coronary angiography confirmed severe calcified lesions (Mintz classification ≥Grade 2), with IVUS unable to pass or showing calcification grade ≥2
* Native coronary artery lesion
* Target vessel diameter 2.5-4.0mm
* Lesion length ≤30mm, suitable for rotational atherectomy
* Clinical indication for PCI: Ischemic cardiomyopathy confirmed by functional testing (e.g., myocardial nuclear scan); Clinical presentation of stable or unstable angina with clear PCI indication
* Planned rotational atherectomy as initial calcium modification technique
* After rotational atherectomy (burr diameter ≤1.5mm), IVUS shows calcification grade still ≥2, or <2 but 2.5mm non-compliant balloon cannot achieve adequate expansion at nominal pressure
* Informed consent signed and agreement to participate in clinical trial
* Able to comply with treatment and complete follow-up

Exclusion Criteria:

* Acute myocardial infarction (AMI) within 7 days, as condition may be unstable and increase periprocedural complication risk
* Target vessel characteristics: Target vessel with thrombus formation, may increase intraoperative embolism risk; Target vessel with chronic total occlusion (CTO), unable to be treated by rotational atherectomy and calcium modification techniques; Target lesion is in-stent restenosis; Target lesion located in coronary artery bypass graft
* Severe heart failure: left ventricular ejection fraction <30%, poor tolerance to PCI surgery, may increase perioperative mortality risk
* Previous treatment history: previous stent implantation or rotational atherectomy in the same target vessel, as complex lesion structure or confounding treatment effects may exist
* Special medical history: Known contrast allergy or severe bleeding tendency (such as active gastrointestinal bleeding), may be unable to tolerate PCI surgery; Patients with other serious comorbidities, expected to be unable to complete 12-month follow-up (such as life expectancy <12 months)
* Pregnancy or lactation: pregnant or lactating women, as intraoperative radiation and drug effects may adversely affect mother and child
* Participation in other clinical trials: patients simultaneously participating in other interventional clinical trials, to avoid mutual influence of different trial intervention measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimum Lumen Diameter (MLD) assessed by intravascular imaging | Immediately post-procedure (within 24 hours after PCI completion)
  The primary efficacy endpoint is the post-procedural minimum lumen diameter (MLD) measured by intravascular imaging (OCT or IVUS) immediately after stent implantation and final post-dilatation. MLD is defined as the smallest luminal diameter within the treated segment. An increase of ≥0.5mm compared to baseline MLD is considered clinically meaningful improvement. The measurement will be performed by the core imaging laboratory using standardized acquisition and analysis protocols with blinded adjudication.

SECONDARY OUTCOMES:
Acute lumen gain assessed by intravascular imaging | Immediately post-procedure (within 24 hours after PCI completion)
  Acute lumen gain is defined as the difference between post-procedural MLD and baseline MLD, measured by OCT or IVUS.
Final stent expansion rate assessed by intravascular imaging | Immediately post-procedure (within 24 hours after PCI completion)
  Stent expansion rate is calculated as the ratio of minimum stent area to the reference vessel area, expressed as a percentage. Assessment includes minimum stent area, stent apposition, and coverage evaluated by OCT/IVUS.
Major Adverse Cardiovascular Events (MACE) at 30 days | 30 days post-procedure
  Composite endpoint of cardiac death, myocardial infarction, and target vessel revascularization at 30 days post-procedure.
Major Adverse Cardiovascular Events (MACE) at 6 months | 6 months post-procedure
  Composite endpoint of cardiac death, myocardial infarction, and target vessel revascularization at 6 months post-procedure.
Major Adverse Cardiovascular Events (MACE) at 12 months | 12 months post-procedure
  Composite endpoint of cardiac death, myocardial infarction, and target vessel revascularization at 12 months post-procedure.
Incidence of periprocedural mechanical complications | During procedure and hospital stay (up to 7 days post-procedure)
  Including coronary perforation (Ellis classification), coronary dissection, acute vessel closure, no-reflow or slow-flow (TIMI flow grade), periprocedural myocardial infarction (Fourth Universal Definition), and acute stent thrombosis (ARC definition).
Bleeding events according to BARC criteria | 30 days post-procedure
  Bleeding events classified according to the Bleeding Academic Research Consortium (BARC) definition, focusing on BARC type 2 or higher bleeding.
Incidence of acute kidney injury | 48-72 hours post-procedure
  Acute kidney injury defined by KDIGO criteria: serum creatinine increase ≥0.3 mg/dL within 48 hours or ≥1.5 times baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zhao, Dr, Principal Investigator — Beijing Chaoyang Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Chaoyang Hospital，Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] Guedeney P, Claessen BE, Mehran R, Mintz GS, Liu M, Sorrentino S, Giustino G, Farhan S, Leon MB, Serruys PW, Smits PC, von Birgelen C, Ali ZA, Genereux P, Redfors B, Madhavan MV, Ben-Yehuda O, Stone GW. Coronary Calcification and Long-Term Outcomes According to Drug-Eluting Stent Generation. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1417-1428. doi: 10.1016/j.jcin.2020.03.053. PMID 32553329
- [Result] Hemetsberger R, Abdelghani M, Toelg R, Mankerious N, Allali A, Garcia-Garcia HM, Windecker S, Lefevre T, Saito S, Slagboom T, Kandzari D, Koolen J, Waksman R, Richardt G. Impact of Coronary Calcification on Clinical Outcomes After Implantation of Newer-Generation Drug-Eluting Stents. J Am Heart Assoc. 2021 Jun 15;10(12):e019815. doi: 10.1161/JAHA.120.019815. Epub 2021 May 29. PMID 34056911
- [Result] De Maria GL, Scarsini R, Banning AP. Management of Calcific Coronary Artery Lesions: Is it Time to Change Our Interventional Therapeutic Approach? JACC Cardiovasc Interv. 2019 Aug 12;12(15):1465-1478. doi: 10.1016/j.jcin.2019.03.038. PMID 31395217